CLINICAL TRIAL: NCT02721511
Title: A Pilot Study to Investigate the Safety and Efficacy of a Novel Furosemide Regimen, Administered Subcutaneously for the Treatment of Fluid Overload and to Evaluate the Feasibility for Home Treatment
Brief Title: A Study to Investigate the Safety and Efficacy of a Novel Furosemide Regimen
Acronym: DIVERSION-HF
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Investigator decision based on new device information.
Sponsor: Todd M Koelling, MD (Other)
Collaborators: scPharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Todd M Koelling, MD, Professor of Internal Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00107057
Record Dates: First submitted 2016-03-17; First posted 2016-03-29 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Acute Decompensated Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Furosemide injection solution 8mg/mL (Experimental): 8mg/mL (total dose=80mg) of furosemide injection solution administered subcutaneously as 30mg over the first hour and then as 12.5 mg per hours over the subsequent 4 hours.
  Interventions: Drug: Furosemide Injection Solution 8mg/mL

INTERVENTIONS:
Drug: Furosemide Injection Solution 8mg/mL — Furosemide Injection Solution, 8 mg/mL, (total dose =80 mg) administered subcutaneously as 30 mg over the first hour and then as 12.5 mg per hour over the subsequent 4 hours by means of the B. Braun Perfusor® Space Infusion Pump System.
  Other Names: SCP-101, Buffered Lasix, Buffered furosemide

SUMMARY:
This is a, prospective, single center, open-label, pilot study to evaluate the safety and efficacy of the subcutaneous administration of a novel furosemide formulation. The results of this pilot study will be reviewed to determine the safety of the subcutaneous treatment regimen and to evaluate patient selection criteria for possible at home treatment. The intent is to conduct a future follow on study looking at the feasibility of at home treatment of patients referred to a hospital for treatment of fluid overload.

DETAILED DESCRIPTION:
In this pilot study, the treatment in the hospital setting will simulate how the patient would be treated at home in the feasibility study. The results of this pilot will be used to inform the design of the feasibility study. The future feasibility study will test the concept that removing the need for professional care for furosemide administration allows a proportion of these patients to go home and be treated safely at home.

A total of 10 patients will be studied using an open label approach to assess efficacy, tolerability and safety of subcutaneous administration of a novel furosemide regimen, administered subcutaneously.

Patients who are referred to the hospital for treatment of fluid overload will complete screening and treatment phases. Subjects meeting the eligibility criteria will be administered a test dose of 80mg furosemide USP administered by intravenous (IV) bolus over 2 minutes. Fluid intake will be restricted during the 2-hour observation period.

Only patients who respond to the test dose of commercially available 80mg intravenous (IV) furosemide (alternatively, bumetanide 2 mg IV ) by means of diuresis in excess of 400 mL over 2 hours will be eligible to enter the treatment phase of the study with the Investigational Medicinal Product. Patients who have responded to the equivalent dose of furosemide or bumetanide as part of their clinical care for heart failure in the hospital within 24 hours of recruitment will not require this test dose and will be eligible for entry into the study provided they meet all of the entry criteria for the study.

Non-responders will be treated in the hospital with usual care.

Investigational Medicinal Product:

Subjects who are Diuretic Responders will be treated with the Investigational Medicinal Product for a period of 24 hours. Furosemide Injection Solution, 8 mg/mL (80 mg total dose) will be administered subcutaneously by means of the B. Braun Perfusor® Space Infusion Pump System. The pump will be programmed to deliver 80mg of furosemide over 5 hours with 30mg administered during the first hour followed by 12.5mg/hour for 4 hours.

Subjects will be treated with twice daily dosing, by default, but may be reduced to once daily if it is desired to reduce the daily urine response. The duration and frequency of the treatment will be determined by the attending cardiologist.

If the subject requires further diuresis after 24 hours, they will be converted to usual care at that time. If the attending cardiologist makes the determination at any time that the diuresis is not adequate, the subject's participation in the study will be stopped, and the patient will convert over to usual care.

Urine output every 24 hours will be recorded, as will daily weights. Serum potassium, sodium, blood urea nitrogen, creatinine and hemoglobin will be assessed daily. All patients will be monitored for heart rhythm continuously during the hospitalization. Temperature every 8 hours will be recorded, and the injection site will be assessed daily for signs of erythema.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male 18 years or older
2. History of heart failure >90-days
3. Presenting to the University of Michigan Health System because of evidence of fluid overload and recommended for admission or observation unit stay to receive intravenous (IV) furosemide therapy.
4. Estimated excess fluid weight of 10 lbs or more from euvolemic state.
5. Estimated jugular venous pressure (JVP) ≥ 10 cm above the right atrium (RA).
6. Evidence of edema up to mid shin or higher
7. Agreeing to sign informed consent and HIPAA authorization
8. Daily dose of furosemide prescribed ≤ 160 mg, or torsemide ≤ 40 mg or bumetanide ≤ 4 mg.

Exclusion Criteria:

1. Pregnant females or women of child-bearing age who are not willing to use an adequate form of contraception
2. Chronic Obstructive Pulmonary Disease (COPD) moderate or worse: FEV1/FCV ratio <0.7 and FEV1 <60 percent predicted.
3. Rapid atrial fibrillation (AF) (HR >100b/min)
4. Hypoxia (resting O2 saturation <9%)
5. Hypotension (systolic blood pressure (SBP) BP < 90 mmHg)
6. Uncontrolled diabetes mellitus (DM) (admission glucose levels > 300 mg/dL)
7. Advanced renal disease (eGFR < 30mL/min/1.73m2)
8. Hypoalbuminemia (Albumin < 3.0 g/dL)
9. Acute coronary syndrome
10. Serum potassium (K+) <3.5 meq/L or using potassium supplements equivalent to > 80meq/day.

13. On experimental medication or currently participating in cardiovascular research study.

14. Urinary tract abnormality or disorder interfering with urination. 15. Allergy to the active and inactive ingredients of the study medication. 16. Inability to comply with study requirements 17. Dementia 18. Ongoing substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2017-03-07 (Actual)

PRIMARY OUTCOMES:
Efficacy endpoint: Urine output per 24 hours | 24 hours
  Efficacy will be measured as the ability of the diuretic regimen given one or two times daily to achieve a net 24 hour urine output of 3000 cc or more over the first 24 hours of the study.
Safety endpoint: Composite of Severe hypokalemia, severe hyperkalemia, moderate to severe worsening of renal function, fever, sepsis, intravenous catheter infection, cardiac dysrhythmia causing syncope or requiring therapy or death | 24 hours
  Safety will be assessed as the composite of developing any of the pre-specified serious adverse events: Severe hypokalemia, severe hyperkalemia, moderate to severe worsening of renal function, fever, sepsis, intravenous catheter infection, cardiac dysrhythmia causing syncope or requiring therapy, death.

SECONDARY OUTCOMES:
Functional Status | 24 hours
  New York Heart Association class
Quality of life | 24 hours
  Kansas City Cardiomyopathy Questionnaire
Congestion Scale | 24 hours
  Change in congestion scale
Breathlessness | 24 hours
  Visual analog scale for dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Todd M Koelling, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States